CLINICAL TRIAL: NCT05248867
Title: A Phase 3, Multicenter Study to Evaluate the Safety and Efficacy of AGN-151586 for the Treatment of Glabellar Lines
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Intramuscular AGN-151586 Injection in Adult Participants With Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M21-500; 2021-003667-10 (EudraCT Number)
Record Dates: First submitted 2022-02-14; First posted 2022-02-21 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; AGN-151586

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received 5 intramuscular injections of placebo in the glabellar complex on Day 1. Based on meeting the retreatment criteria, the participants may have also received 1 open-label treatment of AGN-151586 on Day 43.
  Interventions: Drug: Placebo; Drug: AGN-151586
- AGN-151586 (Experimental): Participants received 5 intramuscular injections of AGN-151586 in the glabellar complex on Day 1. Based on meeting the retreatment criteria, participants may also have received 1 open-label treatment of AGN-151586 on Day 43.
  Interventions: Drug: AGN-151586

INTERVENTIONS:
Drug: Placebo — Placebo solution for injection
  Arms: Placebo
Drug: AGN-151586 — AGN-151586 solution for injection

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. AGN-151586 is an investigational product being developed for the treatment of GL. The purpose of this study was to evaluate the safety and efficacy of AGN-151586 for the treatment of GL in participants with moderate to severe GL.

This was a 12-week study in which eligible subjects were enrolled into the study containing 2 treatment periods, double-blind period and open-label period. Participants were randomly assigned to receive AGN-151586 or placebo. There was 1 in a 4 chance that participants would receive placebo. Around 600 adult participants with moderate to severe GL were to be enrolled in the study in approximately 38 sites across the world.

Participants received either AGN-151586 or Placebo administered as 5 intramuscular injections to the glabellar complex on Day 1. Participants meeting retreatment criteria may have received an open-label treatment of AGN-151586 during the study.

Participants attended regular visits during the study at a study site. The effect of the treatment was checked by medical assessments, blood tests, telephone calls, questionnaires and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to accurately assess their facial lines without the use of eyeglasses (contact lens use is acceptable).
* Participant must have moderate or severe Glabellar Lines at maximum frown as assessed by both the investigator and participant using the Facial Wrinkle Scale (FWS) at Screening and Baseline Day 1 visit.

Exclusion Criteria:

* Uncontrolled systemic disease.
* Presence or history of any medical condition that may place the participant at increased risk following exposure to AGN-151586 or interfere with the study evaluation, including:

  * Diagnosed myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
  * History of facial nerve palsy
  * Infection or dermatological condition at the treatment injection sites
  * Marked facial asymmetry, dermatochalasis, deep dermal scarring, excessively thick sebaceous skin, excessively photodamaged skin, or the inability to substantially lessen facial lines even by physically spreading them apart
  * Any eyebrow or eyelid ptosis at screening or Baseline Day 1 visit as determined by the investigator
* History of known immunization to any botulinum neurotoxin serotype.
* Participants who have reported use of any botulinum neurotoxin of any serotype (including any investigational botulinum neurotoxin product) for aesthetic treatment within the last 6 months prior to Baseline (Day 1 of treatment) and for therapeutic treatment within the last 12 months prior to study drug administration.
* Tattoos, jewelry, or clothing which obscure the glabellar area and cannot be removed.
* Anticipated need for surgery or overnight hospitalization during the study.
* History of surgical procedures on forehead and/or periorbital areas or affecting these areas including any lifting procedure (e.g., rhinoplasty, facial lift, suture lift, thread lift, brow lift, eyelid and/or eyebrow surgery).
* History of periorbital, mid-facial, or upper-facial treatment with semi-permanent or permanent soft tissue fillers (e.g., poly-L-lactic acid, polyalkylimide, polymethylmethacrylate, polytetrafluoroethylene, and silicone), synthetic implantation and/or autologous fat transplantation.
* Known active severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.
* Female participant who is pregnant or breastfeeding, and is considering becoming pregnant or donating eggs during the study or for approximately 30 days after the last dose of study drug or until the end of study, whichever is longer.
* Participant who has been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or is currently enrolled in another clinical study or was previously enrolled in this study.
* Anticipated need for treatment with botulinum neurotoxin of any serotype for any reason during the study (other than study drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (38):
- United States (18):
  - Total Skin and Beauty Derm Ctr /ID# 232378, Birmingham, Alabama
  - Clinical Testing of Beverly Hills /ID# 233195, Encino, California
  - Westside Aesthetics /ID# 232443, Los Angeles, California
  - The Research Center at The Maas Clinic /ID# 241262, San Francisco, California
  - Center for Dermatology and Dermatologic Surgery /ID# 232315, Washington D.C., District of Columbia
  - Steven Fagien MD Aesthetic Eyelid Plastic Surgery /ID# 232439, Boca Raton, Florida
  - Dermatology Clinic & Cosmetic Center /ID# 244295, Baton Rouge, Louisiana
  - Delricht Research /ID# 241253, New Orleans, Louisiana
  - Skincare Physicians /ID# 233938, Chestnut Hill, Massachusetts
  - BOYD Beauty Birmingham /ID# 232383, Birmingham, Michigan
  - Skin Search of Rochester Inc. /ID# 232549, Rochester, New York
  - Aesthetic Solutions /ID# 232389, Chapel Hill, North Carolina
  - Aventiv Research Dublin /ID# 233936, Dublin, Ohio
  - KGL Skin Study Center, LLC /ID# 233549, Newtown Square, Pennsylvania
  - Nashville Center for Laser and Facial Surgery /ID# 242535, Nashville, Tennessee
  - Westlake Dermatology & Cosmetic Surgery - Westlake /ID# 232410, Austin, Texas
  - Dallas Plastic Surgery Institute /ID# 232328, Dallas, Texas
  - Austin Institute for Clinical Research at SBA Dermatology /ID# 232316, Houston, Texas
- Canada (4):
  - Beacon Dermatology Inc /ID# 233227, Calgary, Alberta
  - Alberta DermaSurgery Centre /ID# 241172, Edmonton, Alberta
  - Dr. Wei Jing Loo Medicine Prof /ID# 241863, London, Ontario
  - Erevna Innovations Inc. /ID# 239592, Westmount, Quebec
- Germany (7):
  - Studienzentrum Theatiner46 /ID# 241185, Munich, Bavaria
  - Rosenpark Research /ID# 232391, Darmstadt, Hesse
  - Privatpraxis Dr. Hilton & Partner /ID# 232392, Düsseldorf, North Rhine-Westphalia
  - Noahklinik GmbH /ID# 241184, Kassel
  - Hautok and Hautok-cosmetics /ID# 232393, München
  - Privatpraxis fuer Dermatologie und Aesthetik /ID# 241544, München
  - MediCorium Zentrum fuer Dermatologie und Aesthetik /ID# 241186, Oberursel
- Hungary (4):
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont /ID# 244708, Szeged, Csongrád megye
  - Derm-Surg Kft. /ID# 244709, Kaposvár, Somogy County
  - Derma-B Egeszsegugyi es Szolgaltato Kft. /ID# 244706, Debrecen
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 244707, Pécs
- Poland (5):
  - Instytut Zdrowia Dr Boczarska-Jedynak Sp. Z O.O. Sp.K. /Id# 242990, Oświęcim, Lesser Poland Voivodeship
  - Clinical Research Group Sp. z o.o. /ID# 242988, Warsaw, Masovian Voivodeship
  - High-Med Przychodnia Specjalistyczna /ID# 242973, Warsaw, Masovian Voivodeship
  - Novo-Med Zielinski i Wspolnicy Spolka Jawna /ID# 242986, Katowice, Silesian Voivodeship
  - Dermed Centrum Medyczne Sp. z o.o /ID# 242972, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 638 participants with moderate to severe glabellar lines (GL) at maximum frown were enrolled and randomized in a 3:1 ratio to receive either AGN-151586 or placebo in the Double-blind Period. For those meeting all the retreatment criteria on Day 43, a single open-label treatment with AGN-151586 was administered on the same day.
Groups:
- Placebo/None: Participants received placebo injections during the Double-blind Period but did not meet all the retreatment criteria on Day 43. Participants were followed weekly in the Open-label Period until the Facial Wrinkle Scale (FWS) grades assessed by both investigator and participant returned to moderate or severe (investigator and participant grades did not need to match) before being discontinued from the study after completing either the Early Exit or Study Exit Visit.
- Placebo/AGN-151586: Participants received placebo injections during the Double-blind Period and met all the retreatment criteria on Day 43. A single open-label treatment with AGN-151586 was administered on Day 43. Participants were followed for approximately 6 weeks (through Day 84).
- AGN-151586/None: Participants received AGN-151586 during the Double-blind Period but did not meet all the retreatment criteria on Day 43. Participants were followed weekly in the Open-label Period until the Facial Wrinkle Scale (FWS) grades assessed by both investigator and participant returned to moderate or severe (investigator and participant grades did not need to match) before being discontinued from the study after completing either the Early Exit or Study Exit Visit.
- AGN-151586/AGN-151586: Participants received AGN-151586 during the Double-blind Period and met all the retreatment criteria on Day 43. An additional open-label treatment with AGN-151586 was administered on Day 43. Participants were followed for approximately 6 weeks (through Day 84).
Period: Double-blind Period
Arm/Group | Placebo | AGN-151586 | Placebo/None | Placebo/AGN-151586 | AGN-151586/None | AGN-151586/AGN-151586
Started | 156 | 482 | 0 | 0 | 0 | 0
Completed | 148 | 454 | 0 | 0 | 0 | 0
Not Completed | 8 | 28 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 14 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject due to Adverse Event | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 3 | 8 | 0 | 0 | 0 | 0
Period: Open-label Period
Arm/Group | Placebo | AGN-151586 | Placebo/None | Placebo/AGN-151586 | AGN-151586/None | AGN-151586/AGN-151586
Started | 0 | 0 | 3 | 145 | 17 | 437
Completed | 0 | 0 | 0 | 143 | 0 | 426
Not Completed | 0 | 0 | 3 | 2 | 17 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 1 | 7 | 9
Not completed — Withdrawal by Subject due to Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 5 | 2
Not completed — COVID-19 Infection | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other, not specified | 0 | 0 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat Population: all randomized participants, analyzed according to the treatment groups to which they were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AGN-151586 | Total
Number analyzed (Participants) | 156 | 482 | 638
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (12.48) | 47.1 (12.75) | 47.2 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137 | 429 | 566
  Male | 19 | 53 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 49 | 63
  Not Hispanic or Latino | 142 | 433 | 575
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 16 | 19
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 5 | 21 | 26
  White | 142 | 432 | 574
  More than one race | 3 | 11 | 14
  Unknown or Not Reported | 0 | 0 | 0
Facial Wrinkle Scale (FWS) at Maximum Frown - Participant [Count of Participants; unit: Participants] — Participants' assessment of the severity of glabellar lines (GL) at maximum frown was performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity.
  Participants
    0 = None | 0 | 0 | 0
    1 = Mild | 1 | 3 | 4
    2 = Moderate | 41 | 149 | 190
    3 = Severe | 114 | 330 | 444
Facial Wrinkle Scale (FWS) at Maximum Frown - Investigator [Count of Participants; unit: Participants] — Investigators' assessment of the severity of glabellar lines (GL) at maximum frown was performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity.
  Participants
    0 = None | 0 | 0 | 0
    1 = Mild | 1 | 2 | 3
    2 = Moderate | 41 | 149 | 190
    3 = Severe | 114 | 331 | 445

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Grade 0 or 1 and a ≥ 2-grade Improvement From Baseline on the FWS According to Both Investigator and Subject Assessments of Glabellar Lines (GL) Severity at Maximum Frown at Day 7 [US FDA]
Description: [Primary endpoint for the United States FDA] Percentage of participants achieving a Grade 0 or 1 (none or mild) and a ≥ 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to both investigator and participant assessments of glabellar lines (GL) severity at maximum frown at Day 7 are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Day 7 (Double-blind period)
Population: Intent-to-Treat (ITT) Population: all randomized participants, analyzed according to the treatment groups to which they were randomized. Multiple imputation was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants | 0.6 [0.0 to 1.9] | 60.0 [55.5 to 64.4]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was based on Cochran-Mantel-Haenszel (CMH) test stratified by investigator site, toxin use history (for aesthetic purposes), and baseline Facial Wrinkle Scale score at maximum frown after using multiple imputation for missing data; Rate Difference = 59.3, 95% CI 2-sided [54.7 to 63.9] — Difference: AGN-151586 - Placebo

2. Primary Outcome: Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the FWS According to Participant Assessment of Glabellar Lines (GL) Severity at Maximum Frown at Day 7 [European Union Regulatory Agencies]
Description: [Primary endpoint for European Union regulatory agencies] Percentage of participants with a ≥ 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to participant assessment of glabellar lines (GL) severity at maximum frown at Day 7 are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Day 7 (Double-blind period)
Population: Intent-to-Treat (ITT) Population: all randomized participants, analyzed according to the treatment groups to which they were randomized, with a Baseline Facial Lines Outcome (FLO-11) total score (transformed) of ≤50. Multiple imputation was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 0.8 [0.0 to 2.3] | 61.0 [55.9 to 66.0]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 60.2, 95% CI 2-sided [54.9 to 65.4] — Difference: AGN-151586 - Placebo

3. Primary Outcome: Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the FWS According to Investigator Assessment of Glabellar Lines (GL) Severity at Maximum Frown at Day 7 [European Union Regulatory Agencies]
Description: [Primary endpoint for European Union regulatory agencies] Percentage of participants with a ≥ 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to investigator assessment of glabellar lines (GL) severity at maximum frown at Day 7 are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Day 7 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 0.8 [0.0 to 2.3] | 72.1 [67.5 to 76.7]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 71.4, 95% CI 2-sided [66.5 to 76.2] — Difference: AGN-151586 - Placebo

4. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.
Time Frame: From time of informed consent to end of study; median time on follow-up was 85 days for Double-blind Placebo, AGN-151586, Open-label Placebo/AGN-151586 and AGN-151586/AGN-151586 groups, 50 days for Placebo/None group, and 53 days for AGN-151586/None group
Population: Safety population: all participants who were treated with at least 1 dose of study drug. All safety analyses were performed with participants analyzed by their actual treatment received in the DB period/OL period.
Measure: Number; unit: participants
Groups:
- AGN-151586/None: Participants received AGN-151586 during the Double-blind Period but did not meet all the retreatment criteria on Day 43. Participants were followed weekly in the Open-label Period until the Facial Wrinkle Scale (FWS) grades assessed by both investigator and participant returned to moderate or severe (investigator and] participant grades did not need to match) before being discontinued from the study after completing either the Early Exit or Study Exit Visit.
- AGN-151586/AGN-151586: Participants received AGN-151586 during the Double-blind Period and met all the retreatment criteria on Day 43. A single open-label treatment with AGN-151586 was administered on Day 43. Participants were followed for approximately 6 weeks (through Day 84).
Arm/Group | Placebo | AGN-151586 | Placebo/None | Placebo/AGN-151586 | AGN-151586/None | AGN-151586/AGN-151586
Number analyzed (Participants) | 156 | 482 | 3 | 145 | 17 | 437
participants
  Any TEAE | 44 | 118 | 0 | 32 | 0 | 90
  TESAE | 1 | 3 | 0 | 0 | 0 | 1

5. Secondary Outcome: Percentage of Participants With a Grade 0 or 1 and a ≥ 2-grade Improvement From Baseline on the FWS According to Both Investigator and Participant Assessments of Glabellar Lines (GL) Severity at Maximum Frown Over Time [US FDA]
Description: [Secondary endpoint for the United States FDA] Percentage of participants achieving a Grade 0 or 1 (none or mild) and a ≥ 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to both investigator and participant assessments of glabellar lines (GL) severity at maximum frown over time are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hours 8, 12, 24, 36, and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants
  Hour 8 | 0.0 [0.0 to 0.0] | 7.1 [4.8 to 9.3]
  Hour 12 | 0.6 [0.0 to 1.9] | 15.9 [12.6 to 19.2]
  Hour 24 | 0.6 [0.0 to 1.9] | 30.4 [26.3 to 34.6]
  Hour 36 | 0.6 [0.0 to 1.9] | 43.2 [38.7 to 47.6]
  Hour 48 | 0.6 [0.0 to 1.9] | 50.1 [45.6 to 54.6]
  Day 7 | 0.6 [0.0 to 1.9] | 60.0 [55.5 to 64.4]
  Day 14 | 0.0 [0.0 to 0.0] | 25.3 [21.4 to 29.2]
  Day 21 | 0.0 [0.0 to 0.0] | 2.7 [1.3 to 4.2]
  Day 28 | 0.0 [0.0 to 0.0] | 0.2 [0.0 to 0.6]
  Day 35 | 0.0 [0.0 to 0.0] | 0.4 [0.0 to 1.0]
  Day 43 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

6. Secondary Outcome: Percentage of Participants With a Grade 0 or 1 and a ≥ 2-grade Improvement From Baseline on the FWS According to Investigator Assessment of Glabellar Lines (GL) Severity at Maximum Frown Over Time [US FDA]
Description: [Secondary endpoint for the United States FDA] Percentage of participants with a Grade 0 or 1 (none or mild) and at least a 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to investigator assessment of glabellar lines (GL) severity at maximum frown over time are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hours 8, 12, 24, 36, and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants
  Hour 8 | 1.3 [0.0 to 3.0] | 11.0 [8.2 to 13.8]
  Hour 12 | 0.7 [0.0 to 2.0] | 20.2 [16.6 to 23.8]
  Hour 24 | 0.6 [0.0 to 1.9] | 37.4 [33.1 to 41.8]
  Hour 36 | 0.7 [0.0 to 2.0] | 53.1 [48.6 to 57.6]
  Hour 48 | 0.6 [0.0 to 1.9] | 62.2 [57.9 to 66.6]
  Day 7 | 0.6 [0.0 to 1.9] | 72.6 [68.6 to 76.6]
  Day 14 | 0.0 [0.0 to 0.0] | 32.3 [28.1 to 36.6]
  Day 21 | 0.0 [0.0 to 0.0] | 5.2 [3.2 to 7.3]
  Day 28 | 0.0 [0.0 to 0.0] | 1.3 [0.3 to 2.2]
  Day 35 | 0.0 [0.0 to 0.0] | 0.4 [0.0 to 1.0]
  Day 43 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

7. Secondary Outcome: Percentage of Participants With a Grade 0 or 1 and a ≥ 2-grade Improvement From Baseline on the FWS According to Participant Assessment of Glabellar Lines (GL) Severity at Maximum Frown Over Time [US FDA]
Description: [Secondary endpoint for the United States FDA] Percentage of participants with a Grade 0 or 1 (none or mild) and at least a 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to participant assessment of glabellar lines (GL) severity at maximum frown over time are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hours 8, 12, 24, 36, and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants
  Hour 8 | 0.0 [0.0 to 0.0] | 8.1 [5.7 to 10.5]
  Hour 12 | 0.7 [0.0 to 2.0] | 18.5 [15.0 to 22.0]
  Hour 24 | 0.6 [0.0 to 1.9] | 32.1 [27.9 to 36.3]
  Hour 36 | 0.6 [0.0 to 1.9] | 44.4 [40.0 to 48.9]
  Hour 48 | 1.9 [0.0 to 4.1] | 51.8 [47.3 to 56.3]
  Day 7 | 0.6 [0.0 to 1.9] | 63.3 [58.9 to 67.6]
  Day 14 | 0.0 [0.0 to 0.0] | 29.8 [25.6 to 34.0]
  Day 21 | 0.0 [0.0 to 0.0] | 4.2 [2.4 to 6.1]
  Day 28 | 0.0 [0.0 to 0.0] | 1.9 [0.7 to 3.1]
  Day 35 | 1.3 [0.0 to 3.0] | 1.2 [0.3 to 2.2]
  Day 43 | 0.0 [0.0 to 0.0] | 0.8 [0.0 to 1.7]

8. Secondary Outcome: Percentage of Participants With Achievement of Mostly Satisfied or Very Satisfied on the Facial Lines Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 (Overall Satisfaction) for GL at Day 7 [US FDA]
Description: [Secondary endpoint for the United States FDA] The FLSQ is a validated measure that assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the participant perspective. Participants assessed their overall satisfaction with their glabellar lines using a 5-point verbal descriptor scale (VDS): very dissatisfied, mostly dissatisfied, neither dissatisfied nor satisfied, mostly satisfied, and very satisfied. The percentage of participants mostly satisfied or very satisfied is reported. Percentages are rounded off to nearest single decimal.
Time Frame: Day 7 (Double-blind Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants | 5.1 [1.7 to 8.6] | 77.6 [73.9 to 81.4]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 72.5, 95% CI 2-sided [67.4 to 77.6] — Difference: AGN-151586 - Placebo

9. Secondary Outcome: Percentage of Participants With Achievement of Mostly Satisfied or Very Satisfied on the Facial Lines Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 (Overall Satisfaction) for GL at Hour 24 [United States FDA]
Description: as for outcome 8
Time Frame: Hour 24 (Double-blind Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants | 17.3 [11.4 to 23.2] | 59.2 [54.8 to 63.6]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 41.9, 95% CI 2-sided [34.5 to 49.3] — Difference: AGN-151586 - Placebo

10. Secondary Outcome: Percentage of Participants With Achievement of Mostly Satisfied or Very Satisfied on the Facial Lines Satisfaction Questionnaire (FLSQ) Follow-up Version Item 4 (Natural Look) for GL at Day 7 [US FDA]
Description: [Secondary endpoint for the United States FDA] The FLSQ is a validated measure that assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the participant perspective. Participants assessed their satisfaction with natural look using a 5-point verbal descriptor scale (VDS): very dissatisfied, mostly dissatisfied, neither dissatisfied nor satisfied, mostly satisfied, and very satisfied. The percentage of participants mostly satisfied or very satisfied is reported. Percentages are rounded off to nearest single decimal.
Time Frame: Day 7 (Double-blind Period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 156 | 482
percentage of participants | 9.0 [4.5 to 13.5] | 78.5 [74.8 to 82.2]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 69.5, 95% CI 2-sided [63.7 to 75.3] — Difference: AGN-151586 - Placebo

11. Secondary Outcome: Percentage of Participants With a ≥ 20-point Improvement From Baseline in FLO-11 Total Scores for GL at Day 7 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] The Facial Lines Outcomes (FLO-11) Questionnaire is an 11-item validated measure that assesses appearance-related psychological impacts of glabellar lines (GL) from the participant's perspective. Items 1-10 are assessed on an 11-point numeric rating scale that ranges from 0 (Not at all) to 10 (Very much), with higher scores indicating negative impact. Item 11 is scored in the reverse direction. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Day 7 (Double-blind Period)
Population: Intent-to-Treat (ITT) Population: all randomized participants, analyzed according to the treatment groups to which they were randomized, with a Baseline Facial Lines Outcome (FLO-11) total score (transformed) of ≤50 were included. Multiple imputation was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 8.5 [3.7 to 13.2] | 66.6 [61.8 to 71.5]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 58.2, 95% CI 2-sided [51.3 to 65.0] — Difference: AGN-151586 - Placebo

12. Secondary Outcome: Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the FWS According to Participant Assessment of GL Severity at Maximum Frown at Hour 24 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Percentage of participants with a ≥ 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to participant assessment of glabellar lines (GL) severity at maximum frown at Hour 24 are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hour 24 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 0.8 [0.0 to 2.3] | 30.9 [26.2 to 35.7]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 30.1, 95% CI 2-sided [25.2 to 35.1] — Difference: AGN-151586 - Placebo

13. Secondary Outcome: Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the FWS According to Investigator Assessment of GL Severity at Maximum Frown at Hour 24 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Percentage of participants with a ≥ 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to investigator assessment of glabellar lines (GL) severity at maximum frown at Hour 24 during the Double-Blind Period are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hour 24 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 0.8 [0.0 to 2.3] | 36.5 [31.5 to 41.4]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 35.7, 95% CI 2-sided [30.5 to 40.9] — Difference: AGN-151586 - Placebo

14. Secondary Outcome: Percentage of Participants With a ≥ 1-grade Improvement From Baseline on FWS According to Participant Assessment of GL Severity at Maximum Frown at Hour 24 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Percentage of participants with a ≥ 1-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to participant assessment of glabellar lines (GL) severity at maximum frown at Hour 24 are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hour 24 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 11.5 [6.0 to 17.0] | 64.1 [59.2 to 69.1]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 52.6, 95% CI 2-sided [45.2 to 60.0] — Difference: AGN-151586 - Placebo

15. Secondary Outcome: Percentage of Participants With a ≥ 1-grade Improvement From Baseline on FWS According to Investigator Assessment of GL Severity at Maximum Frown at Hour 24 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Percentage of participants with a ≥ 1-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to investigator assessment of glabellar lines (GL) severity at maximum frown at Hour 24 are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hour 24 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 13.8 [7.9 to 19.8] | 72.5 [67.9 to 77.1]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 58.6, 95% CI 2-sided [51.1 to 66.1] — Difference: AGN-151586 - Placebo

16. Secondary Outcome: Percentage of Participants With Achievement of Mostly Satisfied or Very Satisfied on the Facial Lines Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 (Overall Satisfaction) for GL at Hour 24 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] The FLSQ is a validated measure that assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the participant perspective. Participants assessed their overall satisfaction with their glabellar lines using a 5-point verbal descriptor scale (VDS): very dissatisfied, mostly dissatisfied, neither dissatisfied nor satisfied, mostly satisfied, and very satisfied. The percentage of participants mostly satisfied or very satisfied is reported. Percentages are rounded off to nearest single decimal.
Time Frame: Hour 24 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 16.2 [9.8 to 22.5] | 58.7 [53.6 to 63.7]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 42.5, 95% CI 2-sided [34.4 to 50.6] — Difference: AGN-151586 - Placebo

17. Secondary Outcome: Percentage of Participants With Achievement of Mostly Satisfied or Very Satisfied on the Facial Lines Satisfaction Questionnaire (FLSQ) Follow-up Version Item 4 (Natural Look) for GL at Day 7 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] The FLSQ is a validated measure that assesses treatment expectations, treatment satisfaction, and psychosocial impact of GL from the participant perspective. Participants assessed their satisfaction with natural look using a 5-point verbal descriptor scale (VDS): very dissatisfied, mostly dissatisfied, neither dissatisfied nor satisfied, mostly satisfied, and very satisfied. The percentage of participants mostly satisfied or very satisfied is reported. Percentages are rounded off to nearest single decimal.
Time Frame: Day 7 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants | 7.7 [3.1 to 12.3] | 77.7 [73.3 to 82.0]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 70.0, 95% CI 2-sided [63.7 to 76.3] — Difference: AGN-151586 - Placebo

18. Secondary Outcome: Time to the First ≥ 1-grade Improvement From Baseline on the FWS According to Participant Assessment of GL Severity at Maximum Frown [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Time to the first ≥ 1-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to participant assessment of glabellar lines (GL) severity at maximum frown is reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. For those who did not improve at least 1 grade from Baseline, censoring occurred at the latest visit during the treatment period for which FWS data were available.
Time Frame: From Baseline to Day 43 (Double-blind Period)
Population: Intent-to-Treat (ITT) Population: all randomized participants, analyzed according to the treatment groups to which they were randomized, with a Baseline Facial Lines Outcome (FLO-11) total score (transformed) of ≤50.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
days | 41.9 [0 to 69] | 1.0 [0 to 45]

19. Secondary Outcome: Time to the First ≥1-grade Improvement From Baseline on the FWS According to Investigator Assessment of GL Severity at Maximum Frown [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Time to the first ≥1-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to investigator assessment of glabellar lines (GL) severity at maximum frown is reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. For those who did not improve at least 1 grade from Baseline, censoring occurred at the latest visit during the treatment period for which FWS data were available.
Time Frame: From Baseline to Day 43 (Double-blind Period)
Population: as for outcome 18
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
days | 41.0 [0 to 69] | 0.7 [0 to 45]

20. Secondary Outcome: Percentage of Participants With ≥2-grade Improvement From Baseline on the FWS According to Participant Assessment of GL Severity at Maximum Frown Over Time [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Percentage of participants with at least a 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to participant assessment of glabellar lines (GL) severity at maximum frown over time are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hours 8, 12, 24, 36, and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants
  Hour 8 | 0.0 [0.0 to 0.0] | 7.6 [4.9 to 10.3]
  Hour 12 | 0.8 [0.0 to 2.3] | 17.7 [13.8 to 21.7]
  Hour 24 | 0.8 [0.0 to 2.3] | 30.9 [26.2 to 35.7]
  Hour 36 | 0.8 [0.0 to 2.3] | 44.0 [38.9 to 49.1]
  Hour 48 | 2.3 [0.0 to 4.9] | 50.1 [45.0 to 55.3]
  Day 7 | 0.8 [0.0 to 2.3] | 61.0 [55.9 to 66.0]
  Day 14 | 0.0 [0.0 to 0.0] | 30.5 [25.6 to 35.3]
  Day 21 | 0.0 [0.0 to 0.0] | 4.6 [2.4 to 6.9]
  Day 28 | 0.0 [0.0 to 0.0] | 1.9 [0.5 to 3.3]
  Day 35 | 1.5 [0.0 to 3.7] | 1.4 [0.2 to 2.5]
  Day 43 | 0.0 [0.0 to 0.0] | 0.8 [0.0 to 1.8]

21. Secondary Outcome: Percentage of Participants With ≥2-grade Improvement From Baseline on the FWS According to Investigator Assessment of GL Severity at Maximum Frown Over Time [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Percentage of participants with at least a 2-grade improvement from Baseline on the Facial Wrinkle Scale (FWS) according to investigator assessment of glabellar lines (GL) severity at maximum frown over time are reported. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Hours 8, 12, 24, 36, and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants
  Hour 8 | 1.5 [0.0 to 3.7] | 10.9 [7.7 to 14.1]
  Hour 12 | 0.8 [0.0 to 2.3] | 18.6 [14.5 to 22.6]
  Hour 24 | 0.8 [0.0 to 2.3] | 36.5 [31.5 to 41.4]
  Hour 36 | 0.8 [0.0 to 2.3] | 53.3 [48.1 to 58.4]
  Hour 48 | 0.8 [0.0 to 2.3] | 61.7 [56.6 to 66.7]
  Day 7 | 0.8 [0.0 to 2.3] | 72.1 [67.5 to 76.7]
  Day 14 | 0.0 [0.0 to 0.0] | 32.8 [27.9 to 37.7]
  Day 21 | 0.0 [0.0 to 0.0] | 5.4 [3.0 to 7.7]
  Day 28 | 0.0 [0.0 to 0.0] | 1.1 [0.0 to 2.2]
  Day 35 | 0.0 [0.0 to 0.0] | 0.3 [0.0 to 0.8]
  Day 43 | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]

22. Secondary Outcome: Time to Return to Baseline FWS According to Participant Assessment of FWS at Maximum Frown After Achieving Responder Definition on Day 7 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Time to return to Baseline (Baseline criterion of Moderate or Severe) on the Facial Wrinkle Scale (FWS) according to participant assessment of FWS at maximum frown after achieving responder definition on Day 7 is reported. Responder definition was a rating of None or Mild on the FWS. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. For those who maintained their response, censoring occurred at the latest visit during the treatment period for which FWS was available.
Time Frame: From Baseline to Day 43 (Double-blind Period)
Population: Intent-to-Treat (ITT) Population: all randomized participants, analyzed according to the treatment groups to which they were randomized with a Baseline Facial Lines Outcome (FLO-11) total score (transformed) of ≤50. Participants who did not meet the responder definition on Day 7 were excluded from the analysis; analysis was limited to those that responded.
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 3 | 251
days | 28.0 [15 to 43] | 21.0 [8 to 50]

23. Secondary Outcome: Time to Return to Baseline FWS According to Investigator Assessment of FWS at Maximum Frown After Achieving Responder Definition on Day 7 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] Time to return to Baseline (Baseline criterion of Moderate or Severe) on the Facial Wrinkle Scale (FWS) according to investigator assessment of FWS at maximum frown after achieving responder definition on Day 7 is reported. Responder definition was a rating of None or Mild on the FWS. Assessments were performed using the 4-grade Facial Wrinkle Scale (FWS), where 0=none, 1=mild, 2=moderate, and 3=severe. Higher scores indicate more severity. For those who maintained their response, censoring occurred at the latest visit during the treatment period for which FWS was available.
Time Frame: From Baseline to Day 43 (Double-blind Period)
Population: as for outcome 22
Measure: Median (Full Range); unit: days
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 2 | 280
days | 15.0 [15 to 15] | 21.0 [8 to 50]

24. Secondary Outcome: Percentage of Participants With Achievement of Mostly Satisfied or Very Satisfied on the Facial Lines Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 (Overall Satisfaction) for GL Over Time [European Union Regulatory Agencies]
Description: as for outcome 16
Time Frame: Baseline, Hours 8, 24, and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind Period)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
percentage of participants
  Hour 8 | 14.3 [8.2 to 20.4] | 33.1 [28.3 to 38.0]
  Hour 24 | 16.2 [9.8 to 22.5] | 58.7 [53.6 to 63.7]
  Hour 48 | 8.5 [3.7 to 13.2] | 71.4 [66.7 to 76.0]
  Day 7 | 4.6 [1.0 to 8.3] | 76.9 [72.5 to 81.2]
  Day 14 | 5.8 [1.7 to 10.0] | 69.9 [65.1 to 74.7]
  Day 21 | 2.5 [0.0 to 5.2] | 61.4 [56.3 to 66.5]
  Day 28 | 4.7 [0.9 to 8.4] | 56.1 [50.9 to 61.2]
  Day 35 | 3.8 [0.5 to 7.2] | 58.3 [53.2 to 63.4]
  Day 43 | 4.8 [1.1 to 8.6] | 58.1 [52.9 to 63.4]

25. Secondary Outcome: Percentage of Participants With a ≥ 4-point Improvement From Baseline in FLO-11 Item 10 (Look Angry) for GL at Day 7 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] The Facial Lines Outcomes (FLO-11) Questionnaire is an 11-item validated measure that assesses appearance-related psychological impacts of glabellar lines (GL) from the participant's perspective. Items 1-10 are assessed on an 11-point numeric rating scale that ranges from 0 (Not at all) to 10 (Very much), with higher scores indicating negative impact. Item 11 is scored in the reverse direction. Participants answered FLO-11 Item 10 (Look Angry). Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Day 7 (Double-blind Period)
Population: Intent-to-Treat (ITT) Population: all randomized participants, analyzed according to the treatment groups to which they were randomized, and a Baseline Facial Lines Outcome (FLO-11) total score (transformed) of ≤50. Participants with a score that could improve at least 4 points from Baseline were included. Multiple imputation was used for missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 124 | 353
percentage of participants | 5.6 [1.6 to 9.7] | 54.5 [49.2 to 59.7]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 48.8, 95% CI 2-sided [42.2 to 55.4] — Difference: AGN-151586 - Placebo

26. Secondary Outcome: Percentage of Participants With a ≥ 4-point Improvement From Baseline in FLO-11 Item 5 (Look Less Attractive) for GL at Day 7 [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] The Facial Lines Outcomes (FLO-11) Questionnaire is an 11-item validated measure that assesses appearance-related psychological impacts of glabellar lines (GL) from the participant's perspective. Items 1-10 are assessed on an 11-point numeric rating scale that ranges from 0 (Not at all) to 10 (Very much), with higher scores indicating negative impact. Item 11 is scored in the reverse direction. Participants answered FLO-11 Item 5 (Look Less Attractive). Percentages are rounded off to nearest single decimal.
Time Frame: Baseline, Day 7 (Double-blind Period)
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 128 | 362
percentage of participants | 3.9 [0.5 to 7.3] | 48.1 [42.9 to 53.3]
Statistical Analysis 1: Comparison: Placebo vs AGN-151586; AGN-151586 vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Rate Difference = 44.2, 95% CI 2-sided [38.0 to 50.4] — Difference: AGN-151586 - Placebo

27. Secondary Outcome: Mean Global Assessment of Change in Glabellar Lines (GAC-GL) at Maximum Frown Over Time [European Union Regulatory Agencies]
Description: [Secondary endpoint for European Union regulatory agencies] The GAC-GL Questionnaire assesses the appearance of the participant's GL "now" in comparison with their perspective before treatment. Participants assessed the change in their glabellar lines at maximum frown using a 7-point verbal descriptor scale (VDS): very much improved, much improved, minimally improved, no change, minimally worse, much worse, and very much worse, ranging from 3 to -3. Positive changes indicate improvement, 0 no change, and negative changes indicate worsening.
Time Frame: Hours 24 and 48, Days 7, 14, 21, 28, 35, and 43 (Double-blind Period)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AGN-151586
Number analyzed (Participants) | 130 | 368
units on a scale
  Hour 24 | 0.2 (0.10) | 1.4 (0.07)
  Hour 48 | 0.1 (0.09) | 1.9 (0.06)
  Day 7 | 0.1 (0.08) | 2.2 (0.06)
  Day 14 | 0.1 (0.10) | 1.5 (0.07)
  Day 21 | 0.1 (0.10) | 0.5 (0.07)
  Day 28 | 0.1 (0.10) | 0.2 (0.07)
  Day 35 | 0.1 (0.10) | 0.0 (0.07)
  Day 43 | 0.1 (0.09) | 0.0 (0.06)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the end of the study. The median time on follow-up was 85 days for the Double-blind Placebo and AGN-151586 groups as well as the Open-label Placebo/AGN-151586 and AGN-151586/AGN-151586 groups, 50 days for the Placebo/None group, and 53 days for the AGN-151586/None group.
Arm/Group | Placebo | AGN-151586 | Placebo/None | Placebo/AGN-151586 | AGN-151586/None | AGN-151586/AGN-151586
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/482 | 0/3 | 0/145 | 0/17 | 0/437
Serious Adverse Events (participants affected / at risk) | 1/156 | 3/482 | 0/3 | 0/145 | 0/17 | 1/437
Other Adverse Events (participants affected / at risk) | 9/156 | 31/482 | 0/3 | 8/145 | 0/17 | 14/437
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=156) | AGN-151586 (N=482) | Placebo/None (N=3) | Placebo/AGN-151586 (N=145) | AGN-151586/None (N=17) | AGN-151586/AGN-151586 (N=437)
APPENDICITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=156) | AGN-151586 (N=482) | Placebo/None (N=3) | Placebo/AGN-151586 (N=145) | AGN-151586/None (N=17) | AGN-151586/AGN-151586 (N=437)
HEADACHE (Nervous system disorders) | 9 (10) | 31 (35) | 0 (0) | 8 (8) | 0 (0) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT05248867/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/67/NCT05248867/SAP_001.pdf